CLINICAL TRIAL: NCT02827786
Title: Feasibility of Electromagnetic Acoustic Imaging of Liver Tumours - A Pilot Study
Brief Title: Feasibility of Electromagnetic Acoustic Imaging of Liver Tumours
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Enhanced Medical (Industry)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EMASunnybrook1
Record Dates: First submitted 2016-03-18; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Liver Tumours
Keywords: hepatic tumours
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electromagnetic Acoustic Imaging (Experimental)
  Interventions: Device: Electromagnetic Acoustic Imaging

INTERVENTIONS:
Device: Electromagnetic Acoustic Imaging — Electromagnetic Acoustic imaging (EMA) is a novel experimental platform utilizing the combination of electromagnetic radio frequency (RF) and acoustic waves to enhance ultrasound images. The resultant imaging allows (based on early experimental models) tissue differentiation based on its mechanical and electrical properties. Combined with conventional US scanning, this technology potentially allows high spatial resolution imaging of a target tissue with superimposed high contrast functional information. This is a proof-of-concept pilot study in humans.

SUMMARY:
A single-centre, industry sponsored, proof-of-concept pilot study to assess the feasibility of Electromagnetic Acoustic Imaging (EMA) as an imaging platform in the visualization of hepatic tumours.

DETAILED DESCRIPTION:
STUDY DESIGN Population Single centre pilot study enrolling 30 patients. The study population will comprise of adult patients with documented and characterized focal liver lesion(s) (malignant and/or benign) based on imaging performed at Sunnybrook Health Sciences Centre.

Target lesions and background liver to be studied include:

1. Malignant tumours (metastases (adenocarcinomas and neuroendocrine tumours) and primary hepatic malignancy)
2. Benign tumours (haemangiomas, focal nodular hyperplasia and adenomas)
3. Background liver (remote from target lesion), both normal and fatty liver parenchyma will be included.

Participants must meet the strict inclusion/exclusion criteria for study participation.

Enrollment

1. Patients referred for medical imaging at Sunnybrook Health Sciences Centre and have imaging findings consistent with focal hepatic lesion(s) on conventional US, CECT and/or MRI, characteristic of a specific hepatic tumour (benign or malignant), greater than 1.5cm in size and located within a portion of the liver readily amenable to US assessment. An abdominal radiologist and/or surgical oncologist will identify patients. Recruitment will occur prior to baseline imaging (at time of imaging requisition receipt) or immediately following baseline imaging, either by the study coordinator or surgical oncologist.
2. Patients referred for imaged guided percutaneous biopsy of a focal liver lesion will also be identified and recruited in advance of their biopsy appointment/intervention, either by the study coordinator or referring surgical oncologist (at time of receiving or requesting biopsy respectively).
3. In all cases the responsible physician for the patient will be informed of the intent of the participant, in advance of EMA imaging, thus ensuring recruitment occurs within the circle of care.

Imaging

All EMA imaging will be performed using an investigational EMA device/system, located within the Department of Medical Imaging, Sunnybrook Health Sciences Centre.

Informed consent will be obtained at time of study enrollment, but re-confirmed at time of the EMA study.

Pre-determined target liver lesion(s) (based on baseline diagnostic CT, US or MRI) will be reviewed by an experienced board certified radiologist. Target lesion will be initially evaluated with conventional b-mode US imaging to identify lesion location, size and morphology. Technical feasibility of EMA imaging will be evaluated (imaging window, adequate breath hold etc).

Target lesion will be imaged in two planes (sagittal and transverse) with b-mode, with up to two target lesions assessed per patient. One focal site of background liver parenchyma will also be assessed, remote from the target lesion.

Grey-scale tissue characteristics will be recorded of the target and background parenchyma, including target size, location, and morphology with lesion assigned a conspicuity score by the operator.

EMA imaging will be performed using a dedicated experimental EMA system. Imaging of the pre-determined target lesion(s) and background liver parenchyma will be acquired (see detailed EMA imaging technique below), on a single plane with pre-set region of interest. Qualitative and quantitative parameters will be recorded/stored on the imaging system.

No oral or intravenous contrast agents will be used during this EMA study. Standard or modified ultrasound coupling gel will be used routinely as per standard clinical practice.

Integration with Standard Treatment of Liver Cancer Conventional US together with EMA imaging will be the only additional test/intervention performed as part of this study that are not routinely done for the study population.

Patients will receive standard work-up, treatment and follow-up for their liver lesion(s) according to clinical guidelines and institutional policies. Management and/or treatment will not be modified based on the results of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic liver imaging (US, CT or MRI) prior to enrolment demonstrating characteristic (benign or malignant) focal liver lesion with classic imaging features or focal liver lesion that will undergo histopathological analysis (percutaneous biopsy or surgical resection) following EMA imaging.
2. Focal liver lesion ≥ 1.5cm
3. Pre-determined focal liver lesion in location likely easily visible on US
4. Ability to provide written informed consent to participate in the study

Exclusion Criteria:

1. Pregnant or possibility of pregnancy
2. Cardiac pacemaker implanted cardioverter- defibrillator, neuro-stimulation system, hepatobiliary metallic foreign body or tattoo at proposed site of imaging.
3. Indeterminate focal liver lesion by conventional US, CT and/or MRI imaging and without the prospect of histopathological assessment of lesion(s)
4. Local and/or systemic treatment related to focal liver lesion, prior to EMA imaging.
5. Inability to obtain imaging and/or acceptable quality of grey-scale and/or EMA imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
EMA (colour scale) images will be compared to baseline US grey-scale images for a specific target lesion, as determined by standard of care imaging (US, CT, MRI or PET) and/or histologically proven lesion in a given subject. | 18 months
  EMA (colour scale) images will be compared to baseline US grey-scale images for a specific target lesion, as determined by standard of care imaging (US, CT, MRI or PET) and/or histologically proven lesion in a given subject. EMA colour maps and fused EMA colour with grey-scale US imaging will be assigned a binary outcome for lesion detection (yes/no) and positive results will be graded along a categorical incremental scale with respect to level of EMA signal (i.e. 0 (no signal), 1 (minimal signal), 2 (mild signal) to 5 (good)). Expert readers in diagnostic imaging will obtained outcome measures visually.

SECONDARY OUTCOMES:
US grey-scale and EMA colour maps will be obtained from both target liver lesions and background liver tissue from the same subject and compared. | 18 months
  US grey-scale and EMA colour maps will be obtained from both target liver lesions and background liver tissue from the same subject. Comparison will be made visually for difference in signal (grey-scale and colour respectively) between lesion and background liver. Differences will be assigned a binary classification (yes/no) and graded according level of difference (small, medium or large). Expert readers in diagnostic imaging will obtained outcome measures visually.

CONTACTS AND LOCATIONS:
Overall Officials: Chirag Patel, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No